CLINICAL TRIAL: NCT04119089
Title: Reliability of Gastric Suctioning Compared to Gastric Ultrasound for Residual Gastric Volume Monitoring in Intensive Care Unit Pediatric Patients
Brief Title: Gastric Ultrasound to Monitor Gastric Residual Volume
Acronym: GASTRIPED
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0653
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Mechanical Ventilation Complication; Enteral Feeding Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gastric ultrasound — A first gastric ultrasound will be performed in the supine and the right lateral (RLD) decubitus position, allowing a qualitative analysis of the gastric contents (empty, liquid, solid, solid-liquid). The antral area will also be measured in both positions. The volume of gastric fluid content will be calculated according to the following formula: volume (ml) = -7,8 + (0,035 x antral area in RLD (mm²)) + 0,127 x age (month).
  This examination will be immediately followed by the aspiration of gastric contents through the nasogastric tube used for enteral feeding, into 50-ml syringes, by a nurse blinded to the result of the first ultrasound examination. A second antral ultrasound examination will then be performed, by the same investigator blinded to the volume aspirated.
  The occurrence of regurgitation and / or vomiting occurring within the 12 hours before and after the examination will be recorded.

SUMMARY:
It is currently recommended to start enteral nutrition early in intensive care unit children receiving invasive or non-invasive mechanical ventilation.

Gastrointestinal intolerance is the main complication related to early enteral feeding in intensive care unit patients, characterized by gastroparesis with delayed gastric emptying that may lead to regurgitations, vomiting, pulmonary aspiration, and potentially increased risk of ventilator-associated pneumonia (VAP).

Residual gastric volume (RGV) measurement had been recommended to monitor the tolerance to enteral nutrition in mechanically ventilated patients receiving early enteral feeding.

Nevertheless, several studies have challenged the usefulness of such RGV monitoring, showing that it led to reduced caloric intake without any benefits in terms of reducing the occurrence of vomiting and the incidence of VAP.

This lack of relationship between RGV monitored using gastric suctioning and the occurrence of regurgitation, aspiration and pneumonia may reflect the inaccuracy of the aspiration method used for the measurement of the RGV, as it has been reported in adult patients.

Gastric ultrasonography is a non-invasive and easy-to-use tool allowing accurate preoperative assessment of gastric contents, based on both qualitative examination of the gastric antrum and calculation of gastric content volume. Ultrasound examination of the antrum could therefore constitute an alternative to gastric suctioning for the monitoring of RGV in intensive care unit patients.

This prospective study aims to assess the reliability of the RGV monitoring based on gastric suctioning compared to ultrasound technique. Secondary endpoint is to assess whether increased gastric volume, aspirated or calculated by ultrasound, is an independent risk factor of regurgitation and / or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in intensive care unit, requiring invasive or non-invasive mechanical ventilation for a foreseeable duration > 48 hours.
* Enteral nutrition that has been started for more than 48 hours and less than 7 days.
* Age between 37 weeks of post conceptual age and 18 years.
* Parental consent or consent by the person having parental authority.

Exclusion Criteria:

* Abdominal surgery ≤ 1 year
* History of esophageal, gastric, duodenal, or pancreatic surgery
* Enteral nutrition via jejunostomy or gastrostomy.
* Any situation contraindicating the mobilization of the child in the right lateral decubitus position (uncontrolled hemodynamic instability, unstable neurological injury ...)

Ages: 37 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will be conducted in pediatric intensive care unit patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with an empty stomach after aspiration of gastric contents performed for the residual gastric volume monitoring. | Maximum 1 day (Second gastric ultrasound, performed once aspiration of gastric contents has been achieved)
  Empty stomach is defined as the lack of any gastric content when performing the second gastric ultrasound, after aspiration of gastric contents.

CONTACTS AND LOCATIONS:
Locations (1):
- Service Anesthésie réanimation - Centre Hospitalier Hôpital Femme Mère Enfant Groupement Hospitalier Est - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No